CLINICAL TRIAL: NCT01938885
Title: Hepatic Pseudoaneurysms After Conservatively Managed Liver Injuries
Brief Title: Hepatic Pseudoaneurysms After Trauma
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lene Osterballe, MD, Rigshospitalet, Denmark
Other Study IDs: Lene Osterballe
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Pseudoaneurysm; Abdominal Trauma
MeSH Terms: conditions — Aneurysm, False; Abdominal Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hepatic pseudoaneurysm (HPA) is a rare complication after liver trauma, yet it is potentially fatal, as it can lead to sudden severe haemorrhage. The risk of developing posttraumatic hepatic pseudoaneurysm is one of the reasons why some trauma centres do follow-up CT of patients with liver injuries to take the therapeutic consequence. The aim of this study was to investigate the occurrence of HPA post liver trauma.

ELIGIBILITY:
Inclusion Criteria:

* conservatively managed liver trauma patients with follow-up CT or US

Exclusion Criteria:

* patients who underwent laparotomy because of other intra-abdominal injuries

Ages: 3 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients conservatively managed and radiologically followed-up after liver injury, admitted Trauma Centre at the University hospital of Copenhagen, Rigshospitalet from January 2000 to December 2010.
Sampling Method: Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of hepatic pseudoaneurysm after hepatic trauma | 2000-2010
  All admitted and conservatively treated patients with sustained lever injury due to trauma from 2000-2010 were reviewed in order to investigate the incidence and nature of hepatic pseudoaneurysms after liver trauma

CONTACTS AND LOCATIONS:
Overall Officials: Lene Osterballe, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark